CLINICAL TRIAL: NCT00864006
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Divalproex Sodium 125 MG Delayed Release Tablets Under Fasting Conditions
Brief Title: Bioequivalence Study of Divalproex Sodium 125 MG Delayed Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mitleberg. Ph.D., VP Product Development, Sandoz, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1294
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Valproic Acid

ARMS (2):
- 1 (Experimental): Divalproex Sodium 125 MG Delayed Release Tablets Sandoz
  Interventions: Drug: Divalproex Sodium
- 2 (Active Comparator): Depakote 125 MG DR Tablets Abbott Laboratories USA
  Interventions: Drug: Depakote DR Tablets

INTERVENTIONS:
Drug: Divalproex Sodium
  Arms: 1
Drug: Depakote DR Tablets
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of divalproex sodium 125 MG delayed release tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant findings on physical examination, medical history or laboratory tests on screening

Exclusion Criteria:

* Positive test for HIV or Hepatitis B and C
* History of sensitivity to valproic acid or related compounds

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA Guidelines | 9 Days

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu Chen, MD, Ph.D, FRCP(C), Principal Investigator — Pharma Medica Research, Inc.